CLINICAL TRIAL: NCT03247062
Title: Improving the Quality of Sleep in ICU Patients With a "Sleep Bundle"
Brief Title: Sleep Bundle for Improving Sleep in ICU Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Pr. Bara RICOU, Professor, University Hospital, Geneva
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ICU Sleep - 01
Record Dates: First submitted 2017-05-10; First posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-05

CONDITIONS: Sleep; Intensive Care Unit Syndrome
Keywords: agitation, sleep deprivation, bundle
MeSH Terms: conditions — Psychomotor Agitation; Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: Quality improvement project - before after design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort study (Before-after desgin) (Other): Quality improvement - sleep bundle Intervention consists in a sleep bundle, an aggregate of several propositions to improve the sleep of patients.: implementation of a sleep bundle.
  The entire ICU population will be observed before and after intervention.
  Interventions: Other: Quality improvement - sleep bundle

INTERVENTIONS:
Other: Quality improvement - sleep bundle — implementation of a sleep bundle
  Other Names: A sleep bundle to improve the sleep of patients.

SUMMARY:
Summary of the project :

Lack or disturbances of sleep are major problems in patients staying in intensive care unit (ICU) due to the particular environment. The noises, lack of circadian rhythm of light lead to progressive deafferentation. The patients are then at risk of immune deficiencies, agitation and confusion states, cognitive troubles that may be associated to increased morbidity and mortality in the short and long term. Thus, improvement of the sleep of the ICU patients may impact non only during the ICU stay but also on their future quality of life.

The sleep bundle project is a quality improvement project with a before-after design, consisting in the evaluation of a bundle of measures that may increase the quality and duration of sleep in ICU patients.

The bundle consists in the proposition of eye-mask, ear-plugs, music and/or massage to the patients in parallele to structural and organizational modifications of the service such as the decrease of the alarms sounds, changing the luminosity between day and night, etc.

The principal indicators followed will be:

* The sleep quality of the patients
* The continuous noise intensity in the rooms
* The continuous light intensity in the rooms Baseline - before period: 8 weeks Implementation of the bundle with training of the team: 4 weeks After period: 8 weeks.

DETAILED DESCRIPTION:
Sleep bundle_detailed project _ English

The patients of intensive care unit (ICU) suffer from sleep disorders or lack of sleep due to the particular environment. Among other problems, the noise, the lack of circadian variation of the light lead to a progressive temporal and spatial disorientation. The patients then are subject to a modification of their immunity, present agitation and confusion, neurocognitive disorders with consequences on the morbidity and the short and long-term mortality. An improvement of the sleep of the patients staying in the intensive care will have potentially an impact not only during the stay in the service but also for their future quality of life.

The project " sleep bundle " aims at improving the sleep of the patients by the implementation of a multimodal intervention that consists in a set of measures (or bundle) at different levels: on a structural level in the service), organizational and individual care of the patients.

The intervention, called "sleep bundle" will be proposed to each ICU patient at the bedtime: ear plugs, a mask for eyes, the listening of a soft music, a massage. The whole service structure and organization will be modified by: the installation of a bright light in the daytime and avoidance of light or dark at night, education of the medical and nurse staff in order to increase the awareness of the paitents needs (i.e. limit the light during the night by the use of a shadowless illumination during the night care), a protocol to adapt the volume of the alarms, the implementation of trash cans with shock absorber of lid in every cubicle, the presence of viewable clocks by all the patients (temporal orientation), recalling the necessity of giving to the patients their glasses and hearing aids during daytime.

Design of the project and methodology: this project is a Quality improvement project with the classical BEFORE and AFTER approach. It will measure some quantitative measures and indicators before and after the implementation of the intervention, i.e. the sleep bundle.

Primary objective:

Determine if the sleep of the patients can be improved by the use of one "sleep bundle". The subjective evaluation of the quality of the sleep by the patients will be realized with the "Richard Campbell Sleep Questionnaire (RCSQ)", the analog visual scale, translated into French version, completed by the patient.

The objective evaluation of the depth of the sleep will be realized with the BIS (Index Bispectral), in randomly selected patients according to a table of randomization.

Secondary objectives:

To determine the impact of the implementation of the " sleep bundle " on agitation, delirium, the number of incidents (involuntary removal of naso-gastric tubes, venous lines, endotracheal tubes, etc). The evaluation of the states of agitation and delirium of the patients will be realized via the scores SAS and CAM-ICU.

The following data will be collected in the medical file of patients (SISIF ®):

* Age of the patients, gender, length of ICU stay, history of psychiatric disorders, any dependency (alcohol, benzodiazépines, neuroleptics, tobacco, heroin, methadone, etc).
* Pain scores ( EVA and CPOT), quantity of administered by painkillers, psychotrops, opiates
* Frequency of the care of nursing
* Admission in the room(chamber) during night
* Incidents : involuntary removal of catheters, endotracheal tubes, fall, violence.

The following data will be measured in the environment:

* Luminosity of the cubicle(dock,garage), (the before / later) with a luxmeter
* Monitoring of the noise in the rooms " Soundear Draeger".

The population will consist in:

Inclusion criteria:

* Adults (≥18 years),
* Hospitalized of more than 24 hours in the ICU
* Predictable stay of at least another day
* As soon as the patients is awake, with or without endotracheal tube
* Glasgow ≥12, SAS = 3-4, negative CAM-ICU

Exclusions criteria:

Patients with neurological impairment after medical or surgical insult who require neurological surveillance of more than every 4 hours will not benefit from the sleep bundle.

The sample size was calculated from the average score of RCSQ 49±23 m±DS observed of on 9 experimental patients. We seek to achieve a RCSQ score of ≥65 (with the same DS) in 90 %. 44 patients for the period BEFORE and 44 LATER will be needed. The data of the patients will be collected in a anonymous way.

Every patient holding(retaining) the criteria of inclusion will be included in the project. The estimation practised for the last months before the study period shows that the number of liable patients to be included varies between 5 and 15 patients / week according to the occupation rate of the service.

The duration of 3 periods of the project is going to vary according to the number of patients. By taking into account variations of occupation rate and the possible " drop backs out " according to the clinical evolution of the patient, we plan the next periods:

50 patients during the BEFORE period - duration 8 weeks , 30 patients during the implementation of the bundle-duration 4 weeks, 50 patients AFTER the implementation - duration 8 weeks.

Total duration of the project: 20 weeks.

This project will be sustained in the service thereafter, with a continuous monitoring of the sleep quality of ICU patients (RCSQ ) and some indicators.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 yo),
* Hospitalised for ≥ 24h in ICU
* Planned stay of more than 1 day
* After termination of sedation
* Glasgow ≥ 12, SAS ≥ 3-4, CAM-ICU negative

Exclusion Criteria:

* patients with neueological disease or neurosurgery requiring neurological assessment every 4hours or more

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-02-28 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of the quality of sleep in ICU patients measured by the Richards Campbell Sleep Questionnaire (RCSQ) | 6 months
  Before-after design aiming at increasing the Richards Campbell Sleep Questionnaire (RCSQ) of ICU patients.

SECONDARY OUTCOMES:
agitation episodes | 6 months
  SAS > 6
delirium | 6 months
  CAM ICU +
patient related incident | 6 months
  unvoluntary extubation, cathéters or tube retrieval

IPD SHARING:
Plan to Share IPD: No